CLINICAL TRIAL: NCT00245947
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel- Design, Exploratory Pharmacogenomic, Safety and Activity Study of Orally Administered ERB-041 in Subjects With Inflammation Associated With Active Crohn's Disease
Brief Title: Study Evaluating ERB-041 in Active Crohn's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3142A3-102
Record Dates: First submitted 2005-10-26; First posted 2005-10-28 (Estimated); Last update posted 2009-09-10 (Estimated); Status verified 2009-09

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; Inflammation
MeSH Terms: conditions — Crohn Disease; Inflammation | interventions — ERB 041

INTERVENTIONS:
Drug: ERB-041

SUMMARY:
Evaluate the response of inflammatory serum markers to oral ERB-041 in subjects with inflammation associated with active Crohn's disease.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, minimum 18 years of age with a diagnosis of Crohn's disease greater than 3 months,
* Eligible subjects must have adequate hematologic, renal, and hepatic function.

Other inclusions apply

Exclusion Criteria:

* Use of the following medications within the specified time period before randomization is prohibited:

Within 48 hours before randomization

* Nonsteroidal antiinflammatory drugs (NSAIDs) Within 2 weeks before randomization
* Herbal supplements (except for a daily multivitamin/mineral supplement not containing herbal components).

Other exclusions applies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2004-04; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Inflammatory serum markers
Pharmacogenomics
Safety

SECONDARY OUTCOMES:
Crohn's Disease Activity Index (CDAI) scores.
Cell surface markers
Fecal markers

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer